CLINICAL TRIAL: NCT05434117
Title: Feasibility and Preliminary Efficacy of High-intensity Interval Nordic Walking in Patients With Coronary Artery Disease: A Pilot Randomized Clinical Trial (HIIT-NoW)
Brief Title: Feasibility of High-Intensity Interval Nordic Walking in Patients With Coronary Artery Disease
Acronym: HIIT-NoW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20220260
Record Dates: First submitted 2022-06-14; First posted 2022-06-27 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
Keywords: High-intensity interval training; Nordic walking
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel-group pilot RCT
Who Masked: Outcomes Assessor
Masking Description: Outcome variables will be assessed by study personnel who are blinded to patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval Nordic walking (Experimental): Participants will receive high-intensity interval Nordic walking training.
  Interventions: Behavioral: High-intensity interval Nordic walking
- Control (Active Comparator): Participants will undergo standard cardiovascular rehabilitation.
  Interventions: Behavioral: Standard cardiovascular rehabilitation

INTERVENTIONS:
Behavioral: High-intensity interval Nordic walking — Participants will complete supervised exercise sessions twice weekly for 10 weeks. Exercise specialists will educate participants in proper use of walking poles and basic Nordic walking techniques and supervise the exercise training sessions. HIIT-NoW will be 45 min in duration using Nordic poles and consists of (i) a 10-min warm-up at 30-59% heart rate reserve (HRR, light-to-moderate intensity); (ii) 4 × 4 min of high-intensity work periods at 60-89% HRR (vigorous intensity) interspersed with 3 min of low-intensity work periods at 30-59% HRR (light-to-moderate intensity); and, (iii) a 10-min cooldown at 30-39% HRR (light intensity). To allow participants to acclimatize to the HIIT-NoW protocol, the training intensity will target 60-69% HRR for the first week, 70-79% HRR in the second week, and 80-89% HRR from the third week onward. If participants do not tolerate 89% HRR well, they will exercise as close to 89% HRR as possible.
  Arms: High-intensity interval Nordic walking
Behavioral: Standard cardiovascular rehabilitation — Individuals assigned to standard CR will attend onsite exercise-based CR comprised of one onsite exercise session per week for 8-10 weeks. The onsite CR offers exercise sessions tailored to the fitness of patients and strengthening exercise.
  Arms: Control

SUMMARY:
Coronary revascularization, such as heart bypass surgery (CABG) and percutaneous coronary intervention (PCI [inserting a stent to open up blood vessels]) improve survival for people with coronary artery disease. Yet, many patients suffer from poor physical and mental health after coronary revascularization. Traditional cardiac rehabilitation involving moderate-to-vigorous intensity continuous training (MICT) improves physical and mental health. However, alternative exercise programs, such as high-intensity interval training (HIIT) and Nordic walking may provide superior benefits. Nordic walking is like Nordic skiing but uses specifically designed poles for walking. Nordic walking involved core, upper and lower body muscles, resulting in greater energy expenditure while reducing loading stress at the knee. To date, HIIT used in cardiac rehabilitation settings has focused on lower body (e.g., leg cycling). The investigators are not aware of HIIT protocols that target both upper and lower body at the same time. An exercise program that combines HIIT and Nordic walking (HIIT-NoW) may offer an alternative time-efficient whole-body exercise to improve physical and mental health. This study will test if HIIT-NoW can be an alternative exercise option to improve physical and mental health in patients with coronary artery disease.

DETAILED DESCRIPTION:
Coronary revascularization improves survival for patients with coronary artery disease (CAD). Despite successful coronary revascularization treatment, however, many patients with CAD are left suffering from poor exercise capacity and frequently experience difficulties in performing daily activities (e.g., getting dressed, sitting down or getting up from the toilet) because of diminished cardiovascular function and exercise tolerance. Decreased exercise capacity leads to a dramatic reduction in quality of life (QoL) and more severe depression symptoms. Low exercise capacity, poor quality of life (QoL) and severer depression symptoms heighten the risk of subsequent cardiovascular events and mortality.

Current guidelines recommend that persons with CAD who have undergone coronary artery bypass graft surgery (CABG) or percutaneous coronary intervention (PCI) participate in exercise-based cardiovascular rehabilitation (CR). Exercise-based CR is safe, effective and a class IA recommendation following CABG and PCI. Irrefutable evidence demonstrates that exercise-based CR including moderate-to-vigorous intensity continuous exercise training (MICT) improves exercise capacity, QoL, depression and reduces hospital readmissions and cardiovascular morbidity and mortality. MICT has long been used to manage the physical and mental health of CAD patients as per the Canadian Guidelines for Cardiovascular Rehabilitation and Cardiovascular Disease Prevention; however, such exercise may be less efficient and perceived as less motivating/enjoyable. Growing evidence suggests that non-conventional exercise interventions, such as high-intensity interval training (HIIT) and Nordic walking are more effective exercise modalities, and maybe more enjoyable, to improve clinical outcomes (e.g., exercise capacity, QoL, and depression symptoms) in patients with CAD.

HIIT (repeated bouts of brief high-intensity exercise interspersed with active recovery) is an effective and efficient exercise training paradigm. A recent meta-analysis (n=10 studies) comparing HIIT and MICT in patients with CAD suggests that: (1) HIIT is superior to MICT in improving cardiorespiratory fitness (V̇O2peak) of patients with CAD, an important clinical vital sign and strong predictor of mortality; and, (2) HIIT and MICT are equally effective in improving QoL and depression symptoms in patients including CAD. Increases in cardiorespiratory fitness decrease mortality risk -- every 3.5 ml/kg/min increase in V̇O2peak yields a 13% improvement in survival. Exercise training-induced increases in cardiorespiratory fitness are therefore highly desirable for the improvement of important patient outcomes.

Nordic walking is similar to Nordic skiing but uses specifically designed poles for walking. Nordic walking includes the recruitment of core, upper and lower body muscles, resulting in greater exergy expenditure while reducing loading stress at the knee joint. Regular participation in Nordic walking leads to increased exercise capacity. Although data is limited regarding the impact of Nordic walking in comparison to MICT on mental health in patients with CAD, some studies in patients with heart failure have shown superior improvements in QoL and fewer depressive symptoms following Nordic walking when compared to MICT. Our previous randomized controlled trial simultaneously comparing 12 weeks of supervised HIIT, MICT and Nordic walking in patients with CAD showed that Nordic walking was statistically and clinically superior in increasing functional capacity (i.e., distance walked over 6 minutes), and have similar effects on QoL and depression when compared to HIIT or MICT.

As many adults with cardiovascular disease consider lack of time a barrier to exercise, HIIT may be an appealing exercise training paradigm as cardiovascular health benefits can be achieved in less time when compared to MICT. HIIT may also address other frequently reported deterrents to MICT, including lack of interest and motivation, boredom, not challenging enough, and tailored for older people's needs. To date, HIIT used in CR settings has predominantly focused on lower body (e.g., leg cycling). There are few HIIT protocols that simultaneously target both upper and lower body, such as high-intensity interval Nordic walking (HIIT-NoW). Studies have shown that HIIT and Nordic walking are feasible, enjoyable and have similar or superior effects on physical and mental health when compared to MICT. By combining HIIT and Nordic walking, HIIT-NoW may offer an alternative time-efficient whole-body exercise to improve physical and mental health of patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease treated with PCI or CABG;
* willing to come onsite for exercise sessions;
* able to perform a cardiopulmonary exercise testing (CPET); and,
* at least 40 years of age.

Exclusion Criteria:

* currently participating in a CR program;
* unstable angina or established diagnosis of atrial fibrillation, chronic obstructive pulmonary disease, severe mitral or aortic stenosis, or hypertrophic obstructive cardiomyopathy; or,
* unable to return for 10-week follow-up visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Baseline to week 11 follow up
  Recruitment will be assessed for feasibility. Recruitment will be assessed by the proportion of patients remained interested and randomized after being informed of the requirements of the study
Adherence | Baseline to week 11 follow up
  Adherence will be assessed for feasibility. Adherence will be assessed by the attendance to the prescribed exercise sessions
Compliance | Baseline to week 11 follow up
  Compliance will be assessed for feasibility. Compliance will be assessed by the proportion of participants adhering to prescribed exercise intensity. All HIIT-NoW sessions will be monitored by study personnel and compliance to prescribed exercise intensity will be assessed for each exercise session.
Adverse events | Baseline to week 11 follow up
  Safety will be assessed for feasibility. All mild, moderate, and severe symptoms and adverse events throughout this study will be recorded.
Subjective exercise experiences | Baseline to week 11 follow up
  Subjective exercise experiences will be assessed for feasibility. Physical activity enjoyment will be collected using the PACES.
Self-efficacy | Baseline to week 11 follow up
  Self-efficacy will be assessed for feasibility. Exercise self-efficacy will be assessed using the MSES-R.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Baseline to week 11 follow up
  Cardiorespiratory fitness (V̇O2peak) will be measured by a symptom-limited CPET.
Functional capacity | Baseline to week 11 follow up
  Functional capacity will be assessed by the 6-minute walk test.
Fat mass | Baseline to week 11 follow up
  Fat mass (kg) will be measured using bioelectrical impedance analysis.
Quality of life (QoL) | Baseline to week 11 follow up
  General Quality of life will be assessed using the Medical Outcomes Study Short Form-36. Higher scores indicate better QoL
Heart Disease specific Quality of life (HeartQoL) | Baseline to week 11 follow up
  Heart Disease specific Quality of life (HeartQoL) will be assessed using the disease-specific quality of life questionnaire. Higher scores indicate better HeartQoL (0-3 points).
Depression | Baseline to week 11 follow up
  Depression: will be assessed by the Beck Depression Inventory-II. Higher scores indicate more severe depression symptoms.
Gender | Baseline to week 11 follow up
  Gender: will be assessed using the Genesis-Praxy questionnaire.
Physical activity levels | Baseline to week 11 follow up
  Physical activity levels: Participants will wear a activity monitor (Actigraph GT3X) over the right hip for a week at baseline and follow-up.
Subjective functinal capacity | Baseline to week 11 follow up
  Subjective functional capacity will be assessed by the Duke Activity Status Index questionnaire.
Fat-free mass | Baseline to week 11 follow up
  Fat-free mass (kg) will be measured using bioelectrical impedance analysis.
Waist circumference | Baseline to week 11 follow up
  Waist circumference (cm) will be measured by standardized procedures using a Seca tape measure.
Blood pressure | Baseline to week 11 follow up
  Resting blood pressure will be measured in a seated position after a 5-minute rest period using an automated monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No